CLINICAL TRIAL: NCT00951132
Title: Depression and Cardiovascular Risk Markers: Effects of Rosuvastatin Therapy
Acronym: DECAMERONE
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: Failure to include patients
Sponsor: University Hospital, Akershus (Other)
Collaborators: Oslo University Hospital (Other); AstraZeneca (Industry)
Responsible Party: Principal Investigator, Torbjorn Omland, Professor, University Hospital, Akershus
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: AHUSPP0651
Record Dates: First submitted 2009-08-03; First posted 2009-08-04 (Estimated); Last update posted 2023-02-02 (Actual); Status verified 2023-01

CONDITIONS: Depression
Keywords: Inflammation; Atherosclerosis; Hydroxymethylglutaryl-CoA Reductase Inhibitors
MeSH Terms: conditions — Depression; Inflammation; Atherosclerosis | interventions — Rosuvastatin Calcium

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 2 (Experimental): Rosuvastatin
  Interventions: Drug: rosuvastatin
- 1 (Placebo Comparator): Placebo
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: rosuvastatin — 10mg tablets, once daily in three months
  Arms: 2
Drug: Placebo — tablet, once daily, three months
  Arms: 1

SUMMARY:
The purpose of this study is to investigate whether rosuvastatin decreases measures of inflammation in depressive patients.

DETAILED DESCRIPTION:
Depression is associated with increased risk of cardiovascular disease, in which one possible mechanism is systemic inflammation. Further, patients at high risk of cardiovascular disease, rosuvastatin decreases the risk, especially among patients with increased inflammation. This is a proof-of-concept study to investigate whether the antiinflammatory effect of rosuvastatin is similar in depressive as in patients with cardiovascular disease.

ELIGIBILITY:
Inclusion Criteria:

* Persisting self-reported depressive symptoms > 5 weeks
* Indications of aortic atherosclerosis on PET/CT

Exclusion Criteria:

* Clinical indication of statin use.
* Contraindication of statins, or of PET/CT and MRI.
* Established cardiovascular disease.
* Bipolar disorder og comorbid psychosis.

Ages: 40 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2009-09; Primary Completion 2012-12 (Actual); Study Completion 2013-12 (Actual)

PRIMARY OUTCOMES:
Mean SUV of large arteries | 3 months

SECONDARY OUTCOMES:
Peripheral endothelial function (pulse wave amplitude) | 3 months
Circulatory proinflammatory markers | 3 months
Heart rate variability | 3 months
Depressive symptoms | 3 months

CONTACTS AND LOCATIONS:
Overall Officials: Torbjorn Omland, PhD, Principal Investigator — University Hospital, Akershus
Locations (1):
- Akershus University Hospital, Lorenskog, Akershus, Norway